CLINICAL TRIAL: NCT02490371
Title: The Effectiveness of Combination of Low Frequency Repetitive Transcranial Magnetic Stimulation With Structured Physiotherapy Training Program on Restoring Upper Extremity Function for Patients After Stroke
Brief Title: Adjunct Low Frequency Repetitive Transcranial Magnetic Stimulation With Physiotherapy Enhance Upper Extremity Function Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, HLUKKaYan, Senior Physiotherapist, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT-2015-QEHHK
Record Dates: First submitted 2015-05-31; First posted 2015-07-03 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (1) rTMS- PT Ex Group (Experimental): 1 Hz low frequency rTMS over contra-lesional M1 region for 1200 pulse (20 minutes) at 90% resting motor threshold (rMT) will conduct for 10 consecutive sessions (5 days per week for 2 weeks) and immediately followed by 30- minutes structured physiotherapy upper limb training.
  After the 10 sessions of brain stimulation, the 30-minute structured physiotherapy upper limb training program will continue for another 12 weeks (2 sessions per week)
  Interventions: Device: Low frequency rTMS; Behavioral: structured physiotherapy upper limb training
- (2) Placebo- PT Ex Group (Placebo Comparator): placebo stimulation over contra-lesional M1 region will be conducted for 10 consecutive sessions (5 sessions per week for 2 weeks) of and immediately followed by 30- minutes of structured physiotherapy upper limb training.
  Then, the structured physiotherapy upper limb training will continue for another 12 weeks (2 sessions per week).
  Interventions: Device: Low frequency rTMS; Behavioral: structured physiotherapy upper limb training

INTERVENTIONS:
Device: Low frequency rTMS — 1 Hz low frequency rTMS over contra-lesional M1 region for 1200 pulse at 90% resting motor threshold for 10 sessions.Patients in the rTMS-ex group will receive the experimental rTMS A Magstim Rapid Stimulator (Magstim Company, Whitland, UK) equipped with an air-cooled figure-of-eight coil (each loop 70 mm in diameter) and neuro-navigation system will be used to deliver the intervention.
Behavioral: structured physiotherapy upper limb training — Structural Physiotherapy upper limb training for 30-minutes

SUMMARY:
Stroke is the leading cause of function disability or impairment. Non-promising functional return from upper limb rehabilitation has been reported. With the technology advances, transcranial magnetic stimulation (TMS), which is a form of non-invasive direct brain stimulation, may act as an attenuator in regulating or modulating the cortical excitability in order to facilitate cortical re-organization and enhance behavioral performance. Various therapeutic exercise protocols have been investigated regarding their efficacy in promoting motor recovery of the affected upper limb for patients after stroke and the preliminary results were supportive. However, limited numbers of randomized control clinical trials have been published in investigating the "priming" or "additive" value of low frequency repetitive TMS (rTMS) with combination of structural motor training programs.

Thus the objective of this study is: to determine the effectiveness of the combination of low frequency rTMS on contra-lesional M1 and a structured upper limb motor training program on restoring upper limb function among patients with stroke in sub-acute stage. It is hypothesized that the rTMS, when combined with a structured motor training program, confers additional therapeutic effects on upper limb motor function in subacute stroke patients, when compared with the motor training program alone.

The objectives of this study is to determine the effectiveness of the combination of low frequent rTMS on contra-lesional M1 and a structured upper limb motor training program in restoring upper limb function among patients with subacute stroke.

DETAILED DESCRIPTION:
The proposed study will be a randomized double-blinded controlled trial. 26 stroke patients with upper limb impairment who are receiving the outpatient physiotherapy service at the Queen Elizabeth Hospital and fulfill the eligibility criteria will be recruited and randomized into two interventional groups: (1) rTMS + exercise (rTMS-Ex) group and (2) Placebo rTMS +exercise (Placebo-Ex) group. Both rTMS-Ex and placebo-Ex group will receive 10 consecutive treatment sessions (5 sessions per week), which consists of real rTMS stimulation (rTMS-ex group) or placebo rTMS (placebo-Ex group), followed by 30-minute structured upper limb strengthening and task-specific motor training program. After 2 weeks of brain stimulation and motor training, both groups will continue with the same structured motor training program for another 10 weeks (2 sessions/ week).

1. rTMS-Ex Group 10 consecutive sessions (5 days per week for 2 weeks) of 1 Hz low frequency repetitive transcranial magnetic stimulation over contra-lesional M1 region for 1200 pulse (20 minutes) at 90% motor threshold and immediately followed by 75 minutes structured physiotherapy upper limb training.

   After the 10 sessions of brain stimulation, the 30-minute structured physiotherapy upper limb training program will continue for another 12 weeks (2 sessions per week)
2. Placebo-Ex Group 10 consecutive sessions (5 sessions per week for 2 weeks) of placebo stimulation over contra-lesional M1 region and immediately followed by 30 minutes of structured physiotherapy upper limb training.

Then, the structured physiotherapy upper limb training will continue for another 12 weeks (2 sessions per week).

Evaluation on impairment level, motor performance, physiological measurements and self -perceived disability will be performed at 4 time points: before treatment (T0), immediately after treatment (T1), one-month follow-up (T2) and three-month follow-up (T3). 2-way repeated measures ANOVA will be used to determine whether the rTMS-ex group leads to better outcomes than the placebo-ex group.

ELIGIBILITY:
Inclusion Criteria:

1. First-ever stroke
2. Age >60
3. muscle strength > grade 2 and < grade 5 based on manual muscle testing of hand / fingers of the affected upper limb
4. > 1 month and < 6 months after the onset of stroke

Exclusion Criteria:

1. Substantial cognitive impairment with Mini Mental State Test >24
2. Diagnosis of mental illness
3. Pathological conditions referred to as contra-indications for rTMS in guideline suggested by Wassermann (eg. Cardiac pacemaker, intracranial implants, implanted medication pumps, epilepsy)
4. Unstable cardio-pulmonary conditions -

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ka yan LUK, Principal Investigator — Senior Physiotherapist
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenient sampling method was adopted. Patients who were diagnosed with their first-ever stroke and referred to the Physiotherapy Department at Queen Elizabeth Hospital for post-stroke rehabilitation between November 2015 to December 2016 were screened for eligibility by an independent physiotherapist using inclusion criterias.
Pre-assignment Details: Exclusion criteria:
  1. Mini Mental State Test score ≤ 24;
  2. Mental illness;
  3. Contra-indications to rTMS according to guidelines formulated by Wassermann (e.g., intracranial implants, epilepsy, cardiac pacemaker, implanted medication pumps); 4 Unstable cardio-pulmonary condition.
Groups:
- (1) rTMS- PT Ex Group: 1 Hz low frequency rTMS over contra-lesional M1 region for 1200 pulse (20 minutes) at 90% resting motor threshold (rMT) will conduct for 10 consecutive sessions (5 days per week for 2 weeks) and immediately followed by 30- minutes structured physiotherapy upper limb training.
  After the 10 sessions of brain stimulation, the 30-minute structured physiotherapy upper limb training program will continue for another 12 weeks (2 sessions per week)
  Low frequency rTMS: 1 Hz low frequency rTMS over contra-lesional M1 region for 1200 pulse at 90% resting motor threshold for 10 sessions.Patients in the rTMS-ex group will receive the experimental rTMS A Magstim Rapid Stimulator (Magstim Company, Whitland, UK) equipped with an air-cooled figure-of-eight coil (each loop 70 mm in diameter) and neuro-navigation system will be used to deliver the intervention.
  structured physiotherapy upper limb training: Structural Physiotherapy upper limb training for 30-minutes
- (2) Placebo- PT Ex Group: placebo stimulation over contra-lesional M1 region will be conducted for 10 consecutive sessions (5 sessions per week for 2 weeks) of and immediately followed by 30- minutes of structured physiotherapy upper limb training.
  Then, the structured physiotherapy upper limb training will continue for another 12 weeks (2 sessions per week).
  Low frequency rTMS: 1 Hz low frequency rTMS over contra-lesional M1 region for 1200 pulse at 90% resting motor threshold for 10 sessions.Patients in the rTMS-ex group will receive the experimental rTMS A Magstim Rapid Stimulator (Magstim Company, Whitland, UK) equipped with an air-cooled figure-of-eight coil (each loop 70 mm in diameter) and neuro-navigation system will be used to deliver the intervention.
  structured physiotherapy upper limb training: Structural Physiotherapy upper limb training for 30-minutes
Period: Overall Study
Arm/Group | (1) rTMS- PT Ex Group | (2) Placebo- PT Ex Group
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (1) rTMS- PT Ex Group | (2) Placebo- PT Ex Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (5.8) | 65.1 (3.1) | 66.2 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 12 | 12 | 24
Time since stroke (weeks) [Mean (Standard Deviation); unit: years] | 13.6 (5.8) | 15.1 (7) | 14.3 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change of Cortical Excitability From Baseline to at 4th Weeksand 12th Weeks Training in Motor Evoked Potential at 120% Resting MotorThreshold at Affected Hand
Description: Electromyographic (EMG) activity in first doral interossei measured at 120% resting motor threshold. The motor evoked potential amplitude will be measured peak to peak in millivolt(mV). Higher value mean better control
Time Frame: Baseline and at 4th weeks and at 12th weeks
Measure: Mean (Standard Deviation); unit: millivolt
Groups:
- rTMS Group + Exercise: Patient with rTMS and 30 minutes exercise
- Placebo+ Exercise: Placebo stimulation with exercise
Arm/Group | rTMS Group + Exercise | Placebo+ Exercise
Number analyzed (Participants) | 12 | 12
millivolt
  Baseline | 258.3 (278) | 600 (374.6)
  At 4th week | 323.3 (279.5) | 565 (371.7)
  At 12th week | 369.1 (244.6) | 586 (384.9)

2. Secondary Outcome: Change of Upper Limb Impairment From Baseline to at 4th Weeks & 12 th Weeks Training in Fugl-Meyer Assessment (FM) Scale
Description: Fugl-Meyer Assessment (FM) scale is a stroke-specific, performance-based impairment index, the scale range from 0 to 66.
  25 test items included measurement of movement, coordination, and reflex action of the different parts of the paretic upper extremity. The score could range from 0 to 66. Better motor function was reflected by a higher FMA score
Time Frame: Baseline and at 4th weeks and at 12th weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group + Exercise | Placebo+ Exercise
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 46.7 (13.9) | 48.8 (14.9)
  At 4th week | 52.3 (11.9) | 49.9 (15.3)
  At 12th week | 57.0 (9.6) | 53.3 (16.4)

3. Secondary Outcome: Change of Grip Strength From Baseline to at 4th Weeks and at 12th Weeks Training in Force (Kilogram )
Description: Isometric hand grip strength will be measured using the hand-held dynamometer in kilogram (kg). Higher value reflect better hand grip strength
Time Frame: Baseline and at 4th weeks and at 12th weeks
Measure: Mean (Standard Deviation); unit: kilgograms
Arm/Group | rTMS Group + Exercise | Placebo+ Exercise
Number analyzed (Participants) | 12 | 12
kilgograms
  Baseline | 12.6 (11.3) | 13.8 (10.8)
  At 4th week | 13.9 (10.8) | 13.9 (10.5)
  At 12th week | 15.4 (10.1) | 14.4 (11.1)

4. Secondary Outcome: Change of Upper Limb Function From Baseline to at 4th Weeks Training in Action Research Arm Test (ARAT) Scale
Description: The 19-item Action Research Arm Test has four subscales that assess various aspects of upper limb function (i.e., pinch, grip, grasp, and gross motor). Each item was rated on a 4-point scale from 0 to 3. Scale from 0 to 57.A higher score was indicative of better upper limb function.
Time Frame: Baseline and at 4th weeks and at 12th weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS Group + Exercise | Placebo+ Exercise
Number analyzed (Participants) | 12 | 12
units on a scale
  Baseline | 36.5 (17.8) | 41.1 (17.8)
  At 4th week | 45.4 (11.4) | 41.1 (1.13)
  At 12th week | 51.1 (8.9) | 43.2 (17.9)

5. Secondary Outcome: Change of Reaction Time From Baseline to at 4th Weeks and at 12th Weeks Training in Time Measurement (Seconds)
Description: A simple reaction time will be recorded through a computer system. Time for the patient to reaction to the signal will be measured in seconds (sec). Shorter period of time reflect better reaction time.Lower score means better result
Time Frame: Baseline and at 4th weeks and at 12th weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | rTMS Group + Exercise | Placebo+ Exercise
Number analyzed (Participants) | 12 | 12
seconds
  Baseline | 985.8 (439.9) | 654.2 (285.5)
  At 4th week | 902.2 (398.6) | 651.7 (285.4)
  At 12th week | 837.3 (309.1) | 637.9 (291.2)

6. Secondary Outcome: Change of Health Status Measurement From Baseline to at 4th Weeks and at 12th Weeks in Stroke Impact Scale
Description: The 59-item Stroke Impact Scale (SIS) is a stroke-specific, self-report, health status measure. Total range from 0 to 100. Higher score reflect better result.
Time Frame: Baseline and at 4th & 12 th weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group + Exercise | Placebo+ Exercise
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 59 (13.3) | 65.7 (10.3)
  At 4th week | 64.1 (8.5) | 69.6 (11.2)
  At 12th week | 68.4 (6.9) | 72.7 (11.6)

ADVERSE EVENTS:
Time Frame: Adverse event during the rTMS stimulation , following the whole study period included at 4th weeks up to end of study period at 12th weeks had been reported and recorded.
Description: Headache, seizure
Arm/Group | (1) rTMS- PT Ex Group | (2) Placebo- PT Ex Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (1) rTMS- PT Ex Group (N=12) | (2) Placebo- PT Ex Group (N=12)
seizure (Nervous system disorders) | 0 (0) | 0 (0) — Transcranial magnetic stimulation may casue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT02490371/Prot_SAP_000.pdf